CLINICAL TRIAL: NCT03239535
Title: Allogeneic Mesenchymal Stem Cells for the Critical Limb Ischemia Therapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSC-CLI/FMBA/001
Record Dates: First submitted 2017-07-20; First posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cells (Experimental): Mesenchymal stem cells, Intramuscular injection
  Interventions: Biological: Mesenchymal stem cells
- Normal saline (Placebo Comparator): Normal saline, Intramuscular injection
  Interventions: Biological: Normal saline

INTERVENTIONS:
Biological: Mesenchymal stem cells — Intramuscular injection
  Arms: Mesenchymal stem cells
Biological: Normal saline — Intramuscular injection
  Arms: Normal saline

SUMMARY:
The clinical trial aims to study the safety and efficacy of adult allogeneic mesenchymal stem cells for the treatment of critical limb ischemia.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females in the age group of 18-80 yrs of Caucasian origin.
2. Peripheral artery disease (PAD) against the background of atherosclerosis and diabetes mellitus (DM)
3. Critical lower limb ischemia (stages 3-4 by Fontaine-Pokrovsky or stages 4-6 by Rutherford)
4. Patients with remaining symptoms of critical limb ischemia (CLI) in spite of the performed surgical (endovascular or open) treatment and continuing conservative therapy
5. Patients with absent emergency indications to major amputation
6. Patients planned for the reconstructive surgery with a questionable remote outcome due to compromised blood outflow
7. Ankle Brachial Pressure Index (ABPI) ≤ 0.5 or ankle pressure ≤ 70 mm Hg
8. Patients, if having associated Type II Diabetes, should be on medication and well controlled (HbA1c ≤ 8.5 %)
9. On regular medication for hypertension if needed
10. Normal liver and renal function (or having clinically insignificant deviations, according to the treating physician's opinion)
11. Patients who are able to understand the requirements of the study, and willing to provide voluntary written informed consent, abide by the study requirements, and agree to return for required follow-up visits

Exclusion Criteria:

1. Humid gangrene or acute/chronic infection of lower limb.
2. Dry gangrene with extensive foot lesion (> 1\2).
3. Acute arterial failure.
4. Life-threatening conditions and predicted life expectancy of < 6 months.
5. Presence of neoplasm or bone marrow disease
6. Signs of active or chronic, including latent, haemorrhage
7. Any acute or chronic infectious disease
8. Renal failure determined as twofold or higher elevation of serum creatinine as compared to the upper normal limit
9. Hepatic failure determined as the bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels elevated by two and more times over the upper normal limits
10. Thrombocytopenia (platelet counts < 50,000 /µl), leukocytopenia (WBC < 4,000/µl), immunosuppressive therapy
11. Pronounced neurological deficit
12. Patients with gait disturbance for reasons other than CLI
13. Patients not suitable for cell therapy, by the treating physician's opinion
14. CLI patients requiring amputation at the proximal to the trans-metatarsal level
15. Patients with Type I diabetes
16. Patients having respiratory complications/left ventricular ejection fraction < 25%
17. Stroke or myocardial infarction within last 3 months
18. Patients who are contraindicated for X-ray angiography
19. History of severe alcohol or drug abuse within 3 months of screening
20. Pregnant and lactating women.
21. Patients tested positive for HIV 1, hepatitis C virus (HCV), hepatitis B virus (HBV)
22. Unsigned informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-10-01 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 24 months
  Number of adverse events reported
Amputation-free survival | 24 months
  Number of survived patients

SECONDARY OUTCOMES:
Limb salvage from major amputation | 3, 6, 12, 24 months
  Number of patients who avoided amputation
Relief of the rest pain | Immediate, 3, 6, 12, 24 months
  Rest pain will be measured using the rest pain scale
Improvement in healing trophic disorders | Immediate, 3, 6, 12, 24 months
  Assessment of the severity of trophic ulcers
Improvement in perfusion by the ankle-brachial index | Immediate, 3, 6, 12, 24 months
  Measurements of the ankle-brachial index
Improvement in perfusion by radioisotope scintigraphy | Immediate, 3, 6, 12, 24 months
  Radioisotope scintigraphy study
Improvement in total walking distance (TWD) using a standard treadmill test | Immediate, 3, 6, 12, 24 months
  Standard treadmill test

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir P Baklaushev, MD, PhD, Study Director — Deputy Director; Pavel Yu Orekhov, MD, PhD, Principal Investigator — Vascular Surgeon
Locations (1):
- Federal Research Clinical Center of Federal Medical & Biological Agency, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No